CLINICAL TRIAL: NCT00003309
Title: A Phase II Trial of Preradiation Multiagent Chemotherapy for Adults With "Poor Risk" Medulloblastoma, PNET, and Disseminated Ependymoma
Brief Title: Combination Chemotherapy Plus Radiation Therapy in Treating Adult Patients With Brain Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); SWOG Cancer Research Network (Network)
Responsible Party: Group Chair, Eastern Cooperative Oncology Group
Purpose: Treatment
Other Study IDs: CDR0000066256; E4397; SWOG-E4397
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult medulloblastoma; adult anaplastic ependymoma; adult ependymoma; adult supratentorial primitive neuroectodermal tumor (PNET)
MeSH Terms: conditions — Central Nervous System Neoplasms; Medulloblastoma; Ependymoma | interventions — Filgrastim; Cisplatin; Cyclophosphamide; Etoposide; Vincristine; Chemotherapy, Adjuvant; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: filgrastim
Drug: cisplatin
Drug: cyclophosphamide
Drug: etoposide
Drug: vincristine sulfate
Procedure: adjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining more than one drug and combining chemotherapy with radiation therapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy followed by radiation therapy in treating adult patients with brain cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the complete and partial response rate of patients with adult medulloblastoma, primitive neuroectodermal tumor, or disseminated ependymoma treated with preradiation combination chemotherapy.
* Determine the progression free survival and overall survival of these adult patients treated with combination chemotherapy followed by craniospinal radiation.
* Determine the toxic effects associated with this treatment in these patients.

OUTLINE: Patients receive cisplatin IV over 6 hours, etoposide IV, and vincristine IV over 1-2 minutes on day 1; etoposide IV and cyclophosphamide IV over 1-2 hours on days 2-3; filgrastim (G-CSF) subcutaneously (SC) on days 4-13; and vincristine IV over 1-2 minutes on day 15. Treatment repeats every 42 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.

Within 4-6 weeks after the last chemotherapy course, patients undergo radiotherapy 5 days a week for 6 to 7 weeks.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually for 5-10 years.

PROJECTED ACCRUAL: A total of 33 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed central nervous system cancer including:

  * Medulloblastoma with either local residual disease of greater than 1 cm^2 on MRI following resection or evidence of metastases (M1-4)
  * Other primitive neuroectodermal tumors
  * Ependymoma with evidence of subarachnoid metastases
* Must have less than 1 cm of midline shift or no acute elevated intercranial pressure

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC greater than 4,000/mm^3
* Platelet count greater than 125,000/mm^3
* Hemoglobin greater than 10 g/dL
* No preexisting hematologic condition that would increase toxicity or limit ability to comply with evaluations and follow-up

Hepatic:

* Bilirubin less than 2 times upper limit of normal (ULN)
* SGOT less than 2 times ULN
* Alkaline phosphatase less than 2 times ULN
* No preexisting hepatic condition that would increase toxicity or limit ability to comply with evaluations and follow-up

Renal:

* Creatinine greater than 70 mL/min
* No preexisting renal condition that would increase toxicity or limit ability to comply with evaluations and follow-up

Pulmonary:

* No history of significant pulmonary disease or, if there is preexisting pulmonary disease, then DLCO greater than 60% of predicted
* No preexisting pulmonary condition that would increase toxicity or limit ability to comply with evaluations and follow-up

Other:

* No preexisting psychiatric condition that would increase toxicity or limit ability to comply with evaluations and follow-up
* No prior or concurrent malignancies within the past 5 years except curatively treated carcinoma in situ of the cervix or basal cell or squamous cell skin cancer
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* No increasing doses of steroids for intracranial disease within 3 days of registration

Radiotherapy:

* No prior radiotherapy

Surgery:

* 10-28 days since prior surgical resection OR
* At least 5 days since prior biopsy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 1999-05-04 (Actual); Primary Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul L. Moots, MD, Study Chair — Vanderbilt-Ingram Cancer Center; Larry Kleinberg, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins; Geoffrey R. Barger, MD, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (14):
- United States (14):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Veterans Affairs Medical Center - Lakeside Chicago, Chicago, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Vanderbilt-Ingram Cancer Center at Vanderbilt Medical Center, Nashville, Tennessee
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin

REFERENCES:
- [Result] Moots PL, O'Neill A, Barger GR, et al.: Toxicities associated with chemotherapy followed by craniospinal radiation for adults with poor-risk medulloblastoma/PNET and disseminated ependymoma: a preliminary report of ECOG 4397. [Abstract] J Clin Oncol 22 (Suppl 14): A-1573, 125s, 2004.